CLINICAL TRIAL: NCT06853171
Title: An Open-label, Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of KarXT and Dual-burst Release of Xanomeline With Immediate-release Trospium Chloride in Adolescents With Psychiatric Disorders
Brief Title: Safety, Tolerability, and Pharmacokinetics of KarXT and Dual-burst Release of Xanomeline With Immediate-release Trospium Chloride in Adolescents With Psychiatric Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0022
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: KarXT
- Cohort 2 (Experimental)
  Interventions: Drug: KarXT; Drug: KarX-EC
- Cohort 3 (Experimental)
  Interventions: Drug: KarXT; Drug: KarX-EC

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: Xanomeline and Trospium Chloride Capsule; BMS-986510
Drug: KarX-EC — Specified dose on specified days
  Other Names: Xanomeline Enteric-coated; BMS-986519
  Arms: Cohort 2; Cohort 3

SUMMARY:
This study is designed to assess the safety, tolerability, and pharmacokinetics (PK) of multiple doses and ratios of xanomeline and trospium chloride in an IR capsule (KarXT) and dual-burst release of xanomeline with immediate-release trospium chloride in adolescents with psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* LAR (ie, legal guardian or caregiver) must have signed and dated an IRB/IEC-approved ICF in accordance with regulatory, local, and institutional guidelines.
* Confirmed Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) psychiatric diagnosis of 1 of the following:

  1. Schizophrenia or schizoaffective disorder
  2. Bipolar I or II disorder
  3. Attention-deficit/hyperactivity disorder (ADHD)
  4. Tourette's disorder
  5. Autism spectrum disorder (ASD)
* Participant is judged by the investigator to be clinically stable (eg, no psychiatric hospitalization within the last 6 months; no imminent risk of suicide or injury to self, others, or property).

Exclusion Criteria:

* Any clinically significant neurological, metabolic (including type 1 diabetes), hepatic, renal, hematological, pulmonary, cardiovascular, GI (including active obstructive GI disorders), carcinoma, active biliary disorders (eg, symptomatic gallstones) and/or urological disorder, congestive heart failure (uncontrolled), or CNS infection that would pose a risk to the participants if they were to participate in the study or that might confound the results of the study.
* Participant has a risk for suicidal behavior during the study, as determined by the investigator's clinical judgment and C-SSRS.
* eGFR < 60 mL/min.
* History of Gilbert's Disease or history of liver disease (Child-Pugh class A and higher).
* History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma.
* Participants with history of bladder stones or recurrent UTIs.
* Other protocol defined inclusion/exclusion criteria apply.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Day 43
Number of participants with Serioues AEs (SAEs) | Up to Day 43
Number of participants with AEs of Special Interest (AESIs) | Up to Day 43

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 15
Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) | Up to Day 15
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 15
Time of maximum observed plasma concentration (Tmax) | Up to Day 15
Concentration at the end of a dosing interval (Ctau) | Up to Day 15
Cmax accumulation index (AI_Cmax) | Up to Day 15
  Ratio of maximum observed plasma concentration at steady-state on Day 5 to maximum observed plasma concentration after first dose
AUC accumulation index (AI_AUC) | Up to Day 15
  Ratio of area under the concentration-time curve in 1 dosing interval at steady-state on Day 5 to area under the concentration-time curve in 1 dosing interval after first dose
Ctau accumulation index (AI_Ctau) | Up to Day 15
  Ratio of concentration at the end of the dosing interval at steady-state on Day 5 to maximum observed plasma concentration after first dose
Average concentration within a dosing interval at steady-state (Css-avg) | Up to Day 15
Apparent total body clearance (CLT/F) | Up to Day 15
Effective elimination half-life during dosing interval (T-HALF(eff)) | Up to Day 15
T-HALFeff based on AUC observed (T-HALFeff_AUC) | Up to Day 15
  Effective elimination half-life based on degree of area under the plasma concentration-time curve accumulation observed

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Local Institution - 0005, Little Rock, Arkansas
  - Local Institution - 0006, Orange, California
  - Local Institution - 0007, Decatur, Georgia
  - Local Institution - 0008, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com